CLINICAL TRIAL: NCT03868670
Title: Responsive Neurostimulation For Loss Of Control Eating
Acronym: DBSLOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-46563
Record Dates: First submitted 2019-02-14; First posted 2019-03-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Loss of Control Eating; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Responsive Neurostimulation (Experimental): Surgical arm. Patients expected to receive treatment.
  Interventions: Device: responsive neurostimulation

INTERVENTIONS:
Device: responsive neurostimulation — The RNS® System is a novel, implantable therapeutic device that delivers responsive neurostimulation, an advanced technology designed to continuously monitor brain electrical activity, detect abnormal electrical activity and respond by delivering imperceptible levels of electrical stimulation to normalize that activity before an individual experiences seizures. This is an Early Feasibility Study determining the safety and efficacy of NAc-RNS in the treatment of LOC eating in treatment-refractory obesity.

SUMMARY:
The primary objective of this trial is to assess device function and safety, with secondary objectives including the feasibility.

DETAILED DESCRIPTION:
This is a single site, early feasibility study to support development of a novel therapeutic approach for utilizing the NeuroPace RNS® System for nucleus accumbens responsive neurostimulation (NAc- RNS) to ameliorate loss of control over (LOC) eating in persons with treatment-refractory obesity, specifically those who have failed gastric bypass surgery or sleeve gastrectomy surgery. The primary objectives are to assess the safety & feasibility & potential efficacy of the medical device named the NeuroPace RNS® System.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-60 kg/m2
* Failure of at least one pharmacological agent intended for weight loss or binge eating disorder (select glucagon-like-peptide 1 [GLP-1] receptor agonists for the treatment of type 2 diabetes, which induce clinically meaningful weight loss [i.e., >2% baseline weight], qualify as agents intended for weight loss, as do glucose-dependent insulinotropic polypeptide [GIP]/GLP-1 agonists)
* Failure of at least one form of behavioral therapy, such as weight loss therapy and cognitive behavioral therapy (minimum cumulative trial of 6 months)
* Failure of gastric bypass surgery or sleeve gastrectomy surgery
* Assessment by the study site's bariatric surgeon to rule out technical explanations for suboptimal outcome with an upper GI series within 6 months prior to consent (i.e. a pre-study referral assessment) or prior to surgery during the screening phase.
* Presence of LOC over eating (≥4 LOC episodes per week or ≥16 episodes per month (i.e. 28 days)), as reported on the ELOCS or the EDE interview
* Any medical (including psychiatric) conditions must be monitored actively by appropriate discipline and stable for the past 6 months. Related therapies or medications should be held stable for the study duration.
* Surgical suitability confirmed by a psychiatric examination.
* Subject is able to attend all scheduled clinic appointments on their own or with a caregiver.
* Subject is willing and able to complete signaled EMA assessments.
* Adequate social support (e.g. stable housing, identified family member or close friend as emergency contact) without acute or subacute psychosocial stressors based on screening interview
* Premenopausal women must agree to use acceptable methods of birth control.
* Participants provide voluntary, decisionally capable, and appropriately informed consent. - Subject is able to comply w/ all testing and follow-up requirements defined by the study protocol.
* Participant has no immediate plan for relocation beyond 6 hours of the study site.
* Proficiency with the English language.

Exclusion Criteria:

* Subject has an implanted medical device that delivers electrical energy to the brain.
* Subject has an implantable cardiac pacemaker, defibrillator, or neurostimulator.
* Subject requires diathermy treatments.
* Subject requires transcranial magnetic stimulation (TMS) or electroconvulsive therapy.
* Subject is likely to require repeat magnetic resonance imaging (MRI) after implant of the RNS Neurostimulator and Leads.
* Subject is unable to fit into Computerized Tomography (CT) scanner (500lb upper weight limit for CT scanner).
* Subject is pregnant or intends to become pregnant during the course of the study.
* Subject is participating in a therapeutic investigational drug or device study.
* Subject has medical contraindications for surgery including but not limited to severe cardiovascular, pulmonary, renal, liver, hematological disease, severe coagulopathy, or an acute infectious process.
* Subject has evidence of neurological disorders, e.g. seizure disorder, multiple sclerosis, severe acquired brain injury, severe brain atrophy, subdural hematoma, history of hemorrhagic stroke, or other clinically relevant abnormality on preoperative imaging.
* Subject has a current physical or medical condition that could affect eating behavior (e.g., cancer, pregnancy).
* Subject is actively using medication known to affect eating (e.g., appetite suppressants).
* Subject has a clinically significant or unstable psychiatric condition based on psychiatric screening interview.
* Subject has a clinical diagnosis (past or present) of severe anxiety disorder, severe major depression, psychosis, or anorexia based on diagnostic interview.
* Subject has any lifetime history of suicide attempt, intent or engagement in other forms of self-harm behaviors (e.g. cutting).
* Subject has a history of drug abuse or dependence, including nicotine and alcohol, within the preceding 24 months.
* Subject has current use of alcohol at the rate of > 14 drinks per week or > 4 drinks per occasion or any diagnosis of substance abuse/dependence disorder based on DSM-5.
* There is evidence of incipient dementia or cognitive impairment on Neuropsychological assessment by any score on memory, executive functioning, intellectual functioning, language, or visuospatial domains falling 2SD below the normative mean.
* There is evidence of comprehension difficulties (Token Test <36).
* Subject is unable to provide informed consent to treatment.
* Obesity is secondary to another medical condition, a medication side effect, or a genetic syndrome.
* Subject is a candidate for revision of their bariatric surgery due to anatomical or medical co-morbidities that could be addressed. Of note, revision of a sleeve gastrectomy to a gastric bypass for to reverse weight regain alone is less frequently considered a worthwhile effort as the average weight loss of such a revision is about a 10% weight loss. Thus, patients who have a sleeve and meet the Reinhold classification will be included in this study.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Related Adverse Events [Safety and Tolerability] | 5 years
  Safety of the RNS System and NAc stimulation through evaluation of AE's graded as "related" (vs. not related) to the intervention that will be graded based on severity.
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Count of Participants Exhibiting Overall Decrease in Loss of Control Episodes Per Week | 5 years
  This endpoint will be met if at least 50% of subjects exhibiting a decrease in the number of Loss of Control (LOC) episodes per week. LOC episodes will be assessed by the Eating Loss of Control Scale (ELOCS), a more standardized scale measure and better representation of LOC frequency than the Ecological Momentary Assessment (EMA).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shivacharan RS, Rolle CE, Barbosa DAN, Cunningham TN, Feng A, Johnson ND, Safer DL, Bohon C, Keller C, Buch VP, Parker JJ, Azagury DE, Tass PA, Bhati MT, Malenka RC, Lock JD, Halpern CH. Pilot study of responsive nucleus accumbens deep brain stimulation for loss-of-control eating. Nat Med. 2022 Sep;28(9):1791-1796. doi: 10.1038/s41591-022-01941-w. Epub 2022 Aug 29. PMID 36038628